CLINICAL TRIAL: NCT05242562
Title: Effect of Low-volume (1L) vs Intermediate-volume (2L) Bowel Preparation on Cost-effectiveness and Quality of Life (RESULT Study). A Multicenter Randomized Controlled Trial
Brief Title: Effect of Low-volume (1L) vs Intermediate-volume (2L) Bowel Preparation on Cost-effectiveness and Quality of Life
Acronym: RESULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL79014.091.21
Record Dates: First submitted 2021-09-30; First posted 2022-02-16 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Colonic Polyp
Keywords: colonoscopy; bowel preparation; Quality of life; Costeffectiveness
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Polyethylene Glycols; MoviPrep

STUDY DESIGN:
Intervention Model Description: Patients will be randomized during the pre-colonoscopy hospital visit between a specialized low-volume 1-liter bowel preparation fluid (Pleinvue) or an intermediate-volume 2-liter bowel preparation fluid (Moviprep)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pleinvue (Experimental): a 1L poly ethylene glycol PEG solution with added ascorbate (Pleinvue, Norgine, active ingredients PEG 3350, Sodium ascorbate, Sodium sulfate, Ascorbic acid, Sodium chloride, Potassium chlorid)
  Interventions: Drug: Plenvu
- Moviprep (Active Comparator): a 2L PEG solution with added ascorbate (Moviprep, Norgine, active ingredients Macrogol 3350, Sodium Sulphate Anhydrous, Sodium chloride, Potassium chloride, Ascorbic acid, Sodium ascorbate)
  Interventions: Drug: Moviprep

INTERVENTIONS:
Drug: Plenvu — a recently developed 1 liter bowel preparation fluid that is often used in clinical practice. Patients will receive a split dose protocol, low-residue diet 2 days before colonoscopy, and clear liquid diet 1 day before colonoscopy.
  Other Names: Pleinvue
  Arms: Pleinvue
Drug: Moviprep — a 2 liter widely established 2 liter bowel preparation fluid that is commonly used in clinical practice. Patients will receive a split dose protocol, low-residue diet 2 days before colonoscopy, and clear liquid diet 1 day before colonoscopy.
  Arms: Moviprep

SUMMARY:
Adequate bowel preparation for colonoscopy is paramount for optimal diagnostic accuracy and safety. However, the need for high volumes to clean the colon often makes it difficult for patients to adhere to. Therefore, new low volume bowel preparation fluids have been developed. Little is known on the impact of these low volume bowel preparation fluids (1L), compared to intermediate-volume (2L) laxatives on quality of life (QoL) and cost-effectiveness. This study aims to provide further evidence on the presumed positive effect of ultra-low volume bowel preparation on patients' QoL and cost-effectiveness, in addition to its already demonstrated positive effect on bowel cleansing for colonoscopy.

This multicenter randomized controlled trial (RCT) will be conducted in four hospitals in the Netherlands. Secure web-based questionnaires will be used before starting bowel preparation (baseline, t=0) and within 1 week (t=1) after colonoscopy, to assess the impact of bowel preparation on QoL and explore costs and productivity loss for cost-effectiveness analysis.

DETAILED DESCRIPTION:
Background and aims: Adequate bowel preparation for colonoscopy is paramount for optimal diagnostic accuracy and safety. However, the need for high volumes to clean the colon often makes it difficult for patients to adhere to. Therefore, new low volume bowel preparation fluids have been developed. Little is known on the impact of these low volume bowel preparation fluids (1L), compared to intermediate-volume (2L) laxatives on quality of life (QoL) and cost-effectiveness. This study aims to provide further evidence on the presumed positive effect of ultra-low volume bowel preparation on patients' QoL and cost-effectiveness, in addition to its already demonstrated positive effect on bowel cleansing for colonoscopy.

Study design: This multicenter randomized controlled trial (RCT) will be conducted in four hospitals in the Netherlands. Secure web-based questionnaires will be used before starting bowel preparation (baseline, t=0) and within 1 week (t=1) after colonoscopy, to assess the impact of bowel preparation on QoL and explore costs and productivity loss for cost-effectiveness analysis. Data on colonoscopy findings and complications will be retrieved from the patients' medical record.

Study population: This multicenter study will include 470 patients from 4 hospitals.

Intervention: Patients will be randomized during the pre-colonoscopy hospital visit between a specialized low-volume 1-liter bowel preparation fluid (Pleinvue) or an intermediate-volume 2-liter bowel preparation fluid (Moviprep), which are already both routinely used as bowel preparation for colonoscopy in the Netherlands.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no direct benefit for patients participating in this study. Risk associated with participation are considered minimal, and are limited to the possibility of privacy related issues. Nonetheless, this is considered to be minimal because of the use of pseudonymized data and GDPR compliant databases. In the future, results from this study could possibly benefit patients undergoing colonoscopy, with the possibility of reducing the need for repeat colonoscopies and improving patient experience of colonoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Planned elective colonoscopy for surveillance or diagnostic indications

Exclusion Criteria:

* Therapeutic colonoscopy (e.g. endoscopic mucosal resection (EMR)
* History of (sub) total colectomy
* Inflammatory bowel disease (IBD)
* Inpatient status
* Indication for an intensified bowel preparation regime
* Emergency colonoscopy
* Limited Dutch language skills
* Dementia
* Visual impairment
* Commonly accepted contra-indications for non-iso osmotic bowel preparation and ascorbate:

  * Glucose-6-phosphate-dehydrogenase (G6PD) deficiency
  * (sub)ileus
  * Bowel obstruction or perforation
  * Acute abdomen
  * Gastroparesis
  * intolerance for any of the formulation ingredients
  * Severe renal insufficiency (creatinine clearance < 30mL/min)
  * Congestive heart failure (NYHA III or IV)
  * Phenylketonuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Boston Bowel preparation scale score (total and per segment) | during colonoscopy procedure
  Level of bowel cleanliness achieved with the bowel preparation used. Segmental scores range from 0 to 3, in which 0 is worst and 3 is best. A segmental score of 2 or more is considered adequate for colonoscopy.
Proportion of adequately prepared patients per type of bowel preparation | during colonoscopy procedure
  Level of bowel cleanliness achieved with the bowel preparation used. Segmental boston bowel preparation scores range from 0 to 3, in which 0 is worst and 3 is best. A segmental score of 2 or more is considered adequate for colonoscopy.

SECONDARY OUTCOMES:
absolute score of SF-36 (short-form 36) | within 1 week after colonoscopy, questionnaire 2/2
  Change in scoring on the short-form 36 questionnaire before and after bowel preparation. Higher scores indicate a higher quality of life.
absolute score EQ-5D-5L | within 1 week after colonoscopy, questionnaire 2/2
  Change in scoring on EuroQol group 5Dimension-5Levels questionnaire before and after bowel preparation. Higher scores indicate a higher quality of life.
Correlation of clinical parameters and tolerability to Quality of life scores | questionnaire 2/2, within 1 week after colonoscopy
  Correlation of answers to questionaire on tolerability and relation to bowel cleanliness to scoring on SF-36 (short form 36) and EQ-5D-5L (EuroQol group 5 dimensions 5 levels), higher scores indicate a higher quality of life.
Subgroup differences for absolute scores on SF-36 for colonoscopy indication and prior experience with bowel preparation | questionnaire 2/2, within 1 week after colonoscopy
  Change in QoL scores on SF-36 based on having prior experience with bowel preparation, and differences between colonoscopy indications. SF-36 (short form 36), higher scores indicate a higher quality of life.
Subgroup differences in costs for colonoscopy indication and prior experience with bowel preparation | questionnaire 2/2, within 1 week after colonoscopy
  Change in costs based on having prior experience with bowel preparation, and differences between colonoscopy indications.
Subgroup differences for absolute scores on EQ-5D-5L for colonoscopy indication and prior experience with bowel preparation | questionnaire 2/2, within 1 week after colonoscopy
  Change QoL scores on EQ-5D-5L based on having prior experience with bowel preparation, and differences between colonoscopy indications. EQ-5D-5L (EuroQol group 5 dimensions 5 levels), higher scores indicate a higher quality of life.
Total individual costs | questionnaire 2/2, within 1 week after colonoscopy
  Total costs made per individual for the bowel preparation process, including cost for being absent at work and caregiver costs.
Incremental cost-effectiveness ratio | within 1 week after colonoscopy, questionnaire 2/2
  Change in costs per quality adjusted life years between the low-volume arm and intermediate volume arm.
treating physician advised surveillance interval per study arm | During colonoscopy procedure
  advised surveillance interval correlated to colonoscopy findings and BBPS (boston bowel preparation scale) score by the treating physician. Higher scores indicate higher bowel cleanliness

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The dataset used during this study is available from the corresponding author upon reasonable request
Supporting Information: SAP, CSR, Analytic Code
Time Frame: 15y
Access Criteria: The dataset used during this study is available from the corresponding author upon reasonable request